CLINICAL TRIAL: NCT02604719
Title: Tranexamic Acid and Ethamsylate For Preventing Post Partum Hemorrhage in Patient Undergoing LSCS at High Risk For Post PartumHemorrhage : A Randomized Controlled Trial
Brief Title: Tranexamic Acid and Ethamsylate For Preventing PPH in Patient Undergoing LSCS at High Risk For PPH
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ahmed Alanwar (Other)
Responsible Party: Sponsor-Investigator, Ahmed Alanwar, dr.ahmed alanwar, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TXA&Ethamsylate-PPH
Record Dates: First submitted 2015-11-12; First posted 2015-11-13 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Tranexamic Acid; Ethamsylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tanexamic acid and Ethamsylate (Experimental): 10 ml of the study drugs (1 gm Tranexamic acid and 1 gm Ethamsylate ) slowly (over 30-60 sec ) in the 2 minutes after birth
  Interventions: Drug: Tranexamic Acid and Ethamsylate
- placebo (Placebo Comparator): 10 ml normal saline will be administered intravenously just after birth
  Interventions: Drug: Tranexamic Acid and Ethamsylate

INTERVENTIONS:
Drug: Tranexamic Acid and Ethamsylate — The intervention will be the intravenous administration of 10 ml blinded vial of the study drugs (either 1 gmTranexamic acid and 1 gm Ethamsylate or placebo according to randomization group) slowly (over 30-60 sec ) in the 2 minutes after birth and the routine prophylactic oxytocin and after the cord has been clamped , all generally by the anesthesiologist or obstetrician then a pad will be placed under women buttocks then weighting the pads to allow objective measurement of blood loss.
  Other Names: kapron and dycinon

SUMMARY:
The aim of this study is to compare the effect of low dose of Tranexamic acid (1gm) and Ethamsylate (1gm) after prophylactic oxytocin administration versus placebo with prophylactic oxytocin given in the 2 minutes after child delivery in patient undergoing LSCS at high risk for post partum hemorrhage

DETAILED DESCRIPTION:
Research Question:

Is the combination of Tranexamic acid and Ethamsylate is more effective than oxytocin alone for preventing postpartum hemorrhage if they are given after delivery of the fetus ?

ELIGIBILITY:
Inclusion Criteria:

1. Women undergoing elective caesarean section
2. Patient having one or more risk factor for PPH

   * Multiple pregnancy
   * Polyhydramnios (AFI >25cm)
   * Macrocosmic baby (>4.5 Kg)
   * Prolonged , augmented and obstructed labour
   * Obese patients(BMI >30)
   * Premature rapture of membranes
   * Previous history of PPH
3. Age ≥18 years
4. Gestational Age ≥ 35 Weeks
5. Informed Oral Consent From The Patient

Exclusion Criteria:

1. History of venous thrombosis (DVT and/or Pulmonary embolism) OR arterial thrombosis (angina pectoris , myocardial infarction, stroke)
2. History of epilepsy or seizure
3. Any Known Cardiovascular , renal or liver Disease
4. Autoimmune Diseases
5. Sickle Cell Disease
6. Severe hemorrhagic Disease
7. Placenta Previa.
8. Morbidly adherent Placenta
9. Abruptio placenta
10. Eclampsia, hemolysis, elevated liver enzymes, and low platelet count syndrome
11. Administration Of low molecular weight heparin or Anti platelets the week before delivery .

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-05 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
PPH defined as blood loss ≥500 cc | the first 24hours
  measured by pads placed under women buttocks

SECONDARY OUTCOMES:
severe PPH (>1000 cc), . | first 24 hours